CLINICAL TRIAL: NCT00998478
Title: Cardiovascular Disease Risk Factors and the Effects of a Cross-curricular Physical Activity Intervention in 11-14 Year Olds. Activity Knowledge Circuit
Brief Title: Cardiovascular Disease and the Effects of a Cross-curricular Physical Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glamorgan (Other)
Collaborators: Sports Council Wales (Unknown); University of Wales Institute Cardiff (Unknown)
Responsible Party: Gareth Knox, University of Wales Institute Cardiff
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AKC01
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

ARMS (2):
- Activity prescription (Experimental)
  Interventions: Other: Activity Knowledge Circuits
- Normal Curriculum (No Intervention): Followed normal curriculum including physical education

INTERVENTIONS:
Other: Activity Knowledge Circuits — The activity knowledge circuits were implemented, where in addition to regular physical education (PE) activity was increased by two hours a week over an 18-week period. Participants briskly walked 3200 m twice weekly during curriculum lessons (60 min). Short tasks, in line with current curriculum, were provided by subject teachers for participants to complete at stations set every 400 or 800 m. Crucially participants continued to follow national curriculum whilst exercising. Tasks designed by teachers lasted no longer than 60 seconds at each station. With the exception of PE, each curriculum subject delivered a total of four intervention lessons. Circuits were performed outdoors on school premises, with an indoor course of equal distance used during adverse weather conditions.
  Arms: Activity prescription

SUMMARY:
The purpose of this study is to investigate the effects of a cross-curricular physical activity intervention on cardiovascular disease risk factors in 11-14 year olds. The null hypothesis states that the intervention will have no effect on cardiovascular disease risk factors.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of mortality worldwide. Risk factors associated with cardiovascular disease including obesity, blood pressure and blood lipids have been shown to track from childhood through to adulthood. The prevalence of overweight and obesity for children (4-18 years) in the UK is reported to be 15 % and 4 % respectively. Furthermore, in comparison to England (2.9 %) obesity is more prevalent for those living in Scotland (7.6 %) and Wales (6.5 %). Previous research from two Welsh secondary schools indicate overweight and obesity rates for boys and girls aged 12-13 to be even greater at 26 % and 38 % respectively. Further to this, 19 % were identified as having elevated total cholesterol (≥5.2 mmol/L).

For many, overweight and obesity is the result of the combined effect of excess energy consumption and inadequate physical activity. Previous school-based physical activity interventions have demonstrated modest improvements to cardiovascular disease risk factors by implementing extra-curricular activities or improving current physical education curriculum. Few have attempted to increase physical activity using normally, class-room taught curriculum subjects. This study examines the impact of activity knowledge circuits to combat cardiovascular disease risk factors in 11-14 year old children.

ELIGIBILITY:
Inclusion Criteria:

* Any pupil attending years 7, 8, and 9 of a secondary comprehensive school in South Wales

Exclusion Criteria:

* Any pupil with an injury or illness that prevented them from taking part in any form of physical activity.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease risk factors (obesity, blood pressure, blood lipid & lipoprotein) | 6 Months

SECONDARY OUTCOMES:
Physical activity behaviour and aerobic fitness profile | 6 Months
7 day diet assessment | 6 Months
Maturation status | 6 Months
Motivation to exercise | 6 Months
Psychological well-being, self concept, and cognitive performance | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Gareth J Knox, MSc, Principal Investigator — University of Wales Institute Cardiff
Locations (1):
- Porth County Community School, Porth, Rhondda Cynon Taff, United Kingdom

REFERENCES:
- [Derived] Knox G, Baker JS, Davies B, Faulkner S, Rance J, Rees A, Morgan K, Thomas N. A cross-curricular physical activity intervention to combat cardiovascular disease risk factors in 11-14 year olds: 'activity knowledge circuit'. BMC Public Health. 2009 Dec 15;9:466. doi: 10.1186/1471-2458-9-466. PMID 20003492